CLINICAL TRIAL: NCT03861104
Title: Medikal eğitim Videosu, Septoplasti/Septorinoplasti sonrası Nazal Tampon çekiminde Anksiyetiyi Azaltabilir mi?
Brief Title: Could Medical Educational Video Reduce Anxiety Before Nasal Packing Removal After Septoplasty/Septorhinoplasty?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Pelin Koçdor, Principal Investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KA18/390
Record Dates: First submitted 2019-02-24; First posted 2019-03-04 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Septum Deviated; Septoplasty/Septorhinoplasty
Keywords: septoplasty; nasal packing; anxiety; medical video
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: one group will watch informative video and the control group will not before nasal packing removal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group watched video (Active Comparator): patients will watch the medical video before filling out the spielberger state anxiety inventory at the time of nasal packing removal.
  intervention is watching informative video.
  Interventions: Other: medical educational video
- group without video (No Intervention): patients will fill out the spielberger state anxiety inventory without watching the video at the time of nasal packing removal

INTERVENTIONS:
Other: medical educational video — information based on visual and auditory communication
  Arms: group watched video

SUMMARY:
Septoplasty/septorhinoplasty is one of the most common surgical procedures performed in ENT clinics. Intranasal packing is widely used post-operatively for nasal septum stabilization and bleeding control. Patients experience pain after septoplasty during the removal of nasal packing. These patients may be concerned about pain before nasal packing removal, thus increasing anxiety levels. Various methods are currently employed to reduce this pain. Anxiety is a symptom when a person does not feel safe. Anxiety levels can be objectively measured using different tests including Spielberger state anxiety inventory.

In this digital era, there is a growing tendency to use the popular internet sites as YouTube, Google as a new electronic learning for medical information. The quality of information found on YouTube or other sources could be low and make people more anxious before a minor procedure.

Investigators aim to evaluate the effect of visual and auditory information prepared by the surgeon on anxiety level of patient at nasal packing removal after septoplasty/septorhinoplasty. For this purpose; patients who will undergo septo and septorhinoplasty at Istanbul Baskent University Hospital are recruited. A video of nasal packing removal performed by the surgeon will be watched by the patient and Spielberger state anxiety inventory will be filled out before nasal packing removal. The control group will fill out Spielberger State Anxiety Inventory without watching the video before nasal packing removal. The scores of the groups will be compared and the effect of the video based information on anxiety will be revealed.

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo septoplasty/septorhinoplasty procedures
* patients who will receive nasal packing at their septoplasty septorhinoplasty procedures

Exclusion Criteria:

* patients who will not want to participate to the study
* revision surgeries
* if the patient is taking antidepressants during the last 6 months
* if the patient has a history of a disease that can affect anxiety levels
* if patient wants to be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
The effect of visual and auditory information on anxiety levels by using spielberg state anxiety inventory | 1 year
  The effect of visual and auditory information prepared by the surgeon on anxiety levels at nasal packing removal after septoplasty/septorhinoplasty procedures. Mean score of the inventory is 36-41. The minimum and maximum scores of the inventory are 20 and 80. High score means high anxiety level and low score means low anxiety level.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Hospital, Istanbul, Turkey (Türkiye)